CLINICAL TRIAL: NCT00003778
Title: Phase II Trial of Dolastatin-10 in Patients With Previously Untreated Recurrent/Metastatic Sarcoma
Brief Title: Dolastatin 10 in Treating Patients With Recurrent or Metastatic Soft Tissue Sarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02295; FCCC-98019; NCI-T98-0026; CDR0000066907 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 1999-11-01; First posted 2004-08-27 (Estimated); Last update posted 2013-02-08 (Estimated); Status verified 2000-09

CONDITIONS: Ovarian Cancer; Sarcoma
Keywords: recurrent adult soft tissue sarcoma; stage IV uterine sarcoma; recurrent uterine sarcoma; ovarian sarcoma; stage IV adult soft tissue sarcoma
MeSH Terms: conditions — Ovarian Neoplasms; Sarcoma | interventions — dolastatin 10

ARMS (1):
- Arm I (Experimental): Patients receive dolastatin 10 IV over 10 minutes. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: dolastatin 10

INTERVENTIONS:
Drug: dolastatin 10

SUMMARY:
Phase II trial to study the effectiveness of dolastatin 10 in treating patients who have recurrent or metastatic soft tissue sarcoma. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the response rate in patients with recurrent or metastatic soft tissue sarcomas treated with dolastatin 10.

II. Determine the toxicity of this regimen in this patient population.

OUTLINE: This is an open label, multicenter study. Patients are stratified according to center, prior therapy, histologic subtype, stage of disease at diagnosis, and current status of disease (recurrent vs metastatic).

Patients receive dolastatin 10 IV over 10 minutes. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity.

Patients are followed at 1 month.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven recurrent or metastatic soft tissue sarcoma
* No rhabdomyosarcoma, Ewing's sarcoma, chondrosarcoma, osteogenic sarcoma, mesothelioma, or Kaposi's sarcoma Bidimensionally measurable disease other than previously irradiated disease site(s) even if there has been progression within the radiation field
* Pulmonary nodule(s) at least 1 x 1 cm No brain metastases

PATIENT CHARACTERISTICS:

* Age: 18 and over
* Performance status: ECOG 0 or 1
* Absolute neutrophil count at least 2,000/mm3
* Platelet count at least 100,000/mm3
* Bilirubin no greater than 1.5 mg/dL
* AST and ALT less than 1.5 times upper limit of normal (ULN) (3 times ULN if liver metastases present)
* Creatinine no greater than 1.5 mg/dL
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after study
* No uncontrolled infection
* No history of prior malignancy within the past 5 years except basal cell or squamous cell skin cancer, carcinoma in situ of the cervix, or any other malignancy in complete remission

PRIOR CONCURRENT THERAPY:

* No more than 1 prior chemotherapy regimen in the adjuvant setting
* No prior chemotherapy for metastatic disease
* At least 4 weeks since prior chemotherapy (6 weeks for mitomycin or nitrosoureas)
* At least 4 weeks since prior radiotherapy
* Recovered from prior surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 1999-04; Primary Completion 2000-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Margaret von Mehren, MD, Study Chair — Fox Chase Cancer Center
Locations (4):
- United States (4):
  - University of Colorado Cancer Center, Denver, Colorado
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania